CLINICAL TRIAL: NCT02043353
Title: The Natural History and Outcome of Sleep Disordered Breathing in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-14-RT-03-5510-CTIL
Record Dates: First submitted 2014-01-12; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Winter Vs. Summer: All children that underwent PSG evaluation at the Tel Aviv Medical center between 2005-2010
- Primary snoring: All children that were diagosed with primary snoring at the Tel Aviv Medical center between 2005-2010
- Adenotonsillectomy Vs. Adenoidectomy: All children that underwent adenotonsillectomy or tonsillectomy at the Tel Aviv Medical center between 2005-2008
- repeated PSG: All children that underwent Adenoidectomy / Adenotonsillectomy and two PSG evaluations at the Tel Aviv Medical center between 2005-2012

SUMMARY:
Sleep-disordered breathing in children is characterized by recurrent events of partial or complete upper airway obstruction during sleep, resulting in disruption of normal gas exchange (intermittent hypoxia and hypercapnia) and sleep fragmentation. The major symptom is snoring or noisy breathing. Sleep Disordered Breathing (SDB) is a wide spectrum of disorders that includes primary snoring, UARS and OSA. The main etiology for SDB in children is enlarged tonsils and adenoids and therefore the first line of treatment in pediatric SDB is adenotonsillectomy.

The objectives of this study are:

1. To investigate the natural history of primary snoring
2. To investigate the effect of seasonality on SDB severity
3. To compare the effect of adenoidectomy to adenotonsillectomy in the treatment of SDB in children
4. To characterize the children referred for repeated PSG following adenoidectomy or adenotonsillectomy and the indications for second PSG evaluation.

ELIGIBILITY:
Inclusion Criteria:

* healthy normally developing children that underwent PSG evaluation at the Tel Aviv Medical center between 2005-2010

Exclusion Criteria:

* Chronic medical and neurodevelopmental conditions.
* Congenital anomalies.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Healthy children 0-18 years old that underwent PSG evaluation at the Pediatric Sleep Center at Dana Children's hospital between 2005-2010
Sampling Method: Non-Probability Sample
Enrollment: 2856 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Snoring | 4 years
  Snoring will be assesd by PSQ-Pediatric sleep questionnaire
OSA severity (AHI, mean SpO2, SPo2 nadir) | 4 years
Daytime function | 4 years
  Daytime function will be assesd by PSQ-Pediatric sleep questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel